CLINICAL TRIAL: NCT05301192
Title: Angiotensin-(1-7) Cardiovascular Effects in Aging
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Amy Arnold, Associate Professor of Neural and Behavioral Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY 17401; K99HL159272 (NIH)
Record Dates: First submitted 2022-03-17; First posted 2022-03-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Aging
Keywords: cardiovascular; blood pressure; autonomic nervous system; renin-angiotensin system; endothelial
MeSH Terms: interventions — angiotensin I (1-7); Acetates; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Angiotensin-(1-7) (Experimental): Participants will receive intravenous angiotensin-(1-7) at one study visit for 110 minutes. Angiotensin-(1-7) will be given in escalating doses of 2 ng/kg/min, 4 ng/kg/min, and 8 ng/kg/min. Each of these doses will be infused for 10 minutes. Following the dose escalation, angiotensin-(1-7) will be given at 8 ng/kg/min for an additional 80 minutes. Infusion rates will be calculated for each participant based on body mass.
  Interventions: Drug: Angiotensin-(1-7)
- Saline (Placebo Comparator): Participants will receive intravenous saline at one study visit for 110 minutes total. The volume of saline will match the volume of angiotensin-(1-7) infused. Infusion rates will be calculated for each participant based on body mass.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin-(1-7) — This is a biologically active endogenous angiotensin peptide that may play an important role in regulation of blood pressure.
  Other Names: Angiotensin I/II (1-7) Acetate
  Arms: Angiotensin-(1-7)
Drug: Saline — Saline will be used as the placebo comparator.
  Other Names: Normal saline; 0.9% sodium chloride
  Arms: Saline

SUMMARY:
Aging is an independent risk factor for developing hypertension and cardiovascular disease; however, the mechanisms underlying age-related cardiovascular disease remain poorly understood. One hallmark of aging is an increase in sympathetic nervous system activity, which can decrease the number and/or sensitivity of β2 adrenergic receptors to reduce dilation of blood vessels and increase blood pressure. Identifying new targets to restore vascular β2 adrenergic receptor signaling may help reduce cardiovascular risk in aging. This study will test the hypothesis that angiotensin-(1-7), a protective hormone of the renin-angiotensin system, can reduce cardiovascular sympathetic outflow and blood pressure and improve endothelial function in older healthy humans.

DETAILED DESCRIPTION:
A randomized, double blind, placebo-controlled, crossover study will be conducted to determine if acute intravenous angiotensin-(1-7) infusion can reduce cardiovascular sympathetic tone and blood pressure and improve the function of blood vessels in older healthy individuals. This is an outpatient study that requires a screening visit, and if eligible, two study visits separated by at least one week in the Clinical Research Center within the Penn State Milton S. Hershey Medical Center. The study visits will include intravenous infusion of angiotensin-(1-7) or saline for approximately two hours, starting with increasing doses and holding at a steady-state dose. Endothelial function will be measured and blood samples and endothelial cells collected at baseline and at the end of infusions. Blood pressure, heart rate, and muscle sympathetic nerve activity via microneurography will be measured throughout the study. Each study visit will last approximately 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all races and ethnicities
* Capable of giving informed consent
* Fluent in written and spoken English
* Age 65-80 years
* Body mass index (BMI) between 18.5 and 30 kg/m2
* Normotensive defined as seated blood pressure <130/80 mmHg and without hypertensive medications
* Satisfactory history and physical exam

Exclusion Criteria:

* Age < 65 or > 80 years
* Women who are pregnant, nursing, or taking hormone replacement therapy
* Decisional impairment
* Prisoners
* Current or recent (less than 6 months) recreational drug history or excessive alcohol abuse history (greater than 14 drinks per week)
* Current smokers
* Highly trained athletes
* Evidence of type I or type II diabetes (fasting glucose > 126 mg/dL or use of anti-diabetic medications)
* Hypertension or history of serious cardiovascular disease (e.g., myocardial infarction within 6 months, symptomatic coronary artery disease, presence of angina pectoris, significant arrhythmia, congestive heart failure, deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, hypertrophic cardiomyopathy) or cerebrovascular disease (e.g., cerebral hemorrhage, stroke, transient ischemic attack).
* History or presence of immunological or hematological disorders
* Impaired hepatic function [aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels >2 times upper limit of normal range]
* Impaired renal function (serum creatinine >2.0 mg/dl)
* Anemia
* Taking drugs known to influence sympathetic activity (e.g. serotonin-norepinephrine reuptake inhibitors, norepinephrine transporter inhibitors, stimulants).
* Treatment with anticoagulants (e.g. warfarin)
* Treatment with chronic systemic glucocorticoid therapy (>7 consecutive days in 1 month in the 1-month preceding the study)
* Treatment with any investigational drug in the 1-month preceding the study
* Known allergy or contraindication to angiotensin converting enzyme inhibitors or angiotensin receptor blockers, both of which increase endogenous angiotensin-(1-7) levels as part of their mechanism of action
* Inability to give, or withdraw, informed consent

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Sympathetic Nerve Burst Rate | 110 minutes
  Muscle sympathetic nerve burst rate will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.

SECONDARY OUTCOMES:
Change in Muscle Sympathetic Nerve Burst Incidence | 110 minutes
  Muscle sympathetic nerve burst incidence will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.
Change in Muscle Sympathetic Nerve Amplitude | 110 minutes
  Muscle sympathetic nerve amplitude will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.
Change in Muscle Sympathetic Nerve Total Activity | 110 minutes
  Muscle sympathetic nerve total activity will be measured continuously using peroneal nerve microneurography during angiotensin-(1-7) versus saline infusion.
Change in Brachial Artery Diameter | 110 minutes
  A blood pressure cuff will be inflated to a suprasystolic pressure for 5 minutes then deflated. Brachial artery diameter will be measured continuously before, during, and after cuff inflation using duplex ultrasound at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Systolic and Diastolic Blood Pressure | 110 minutes
  Blood pressure will be measured continuously with a finger and arm cuff during angiotensin-(1-7) versus saline infusion.
Change in Heart Rate | 110 minutes
  Heart rate will be measured continuously by electrocardiogram during angiotensin-(1-7) versus saline infusion.
Change in Heart Rate Variability | 110 minutes
  Heart rate variability will be calculated from the continuous electrocardiogram recordings obtained during angiotensin-(1-7) versus saline infusion.
Change in Plasma Catecholamines | 110 minutes
  Circulating catecholamine levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.

OTHER OUTCOMES:
Change in Angiotensin II | 110 minutes
  Plasma angiotensin II levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Angiotensin-(1-7) | 110 minutes
  Plasma angiotensin-(1-7) levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Renin Activity | 110 minutes
  Plasma renin activity will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.
Change in Aldosterone | 110 minutes
  Plasma or serum aldosterone levels will be measured in blood samples obtained at baseline and at the end of angiotensin-(1-7) versus saline infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Arnold, PhD, Principal Investigator — Pennsylvania State University College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No